CLINICAL TRIAL: NCT01198821
Title: A Phase I Study of Oral Sodium Bicarbonate in Patients With Unresectable Pancreatic Carcinoma Treated With Gemcitabine
Brief Title: Gem-TABS in Unresectable Pancreatic Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Reliable Cancer Therapies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16123
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Pancreatic Cancer
Keywords: pancreas; adenocarcinoma; metastatic; unresectable
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma; Neoplasm Metastasis | interventions — Sodium Bicarbonate; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral sodium bicarbonate and Gemcitabine (Experimental)
  Interventions: Drug: Sodium bicarbonate (g/kg/day); Drug: Gemcitabine (mg/m²)

INTERVENTIONS:
Drug: Sodium bicarbonate (g/kg/day) — Dose Escalation - Level 1: 0.3, Level 2: 0.5, Level 3: 0/7, Level 4: 1.0
Drug: Gemcitabine (mg/m²) — Dose Escalation - Level 1: 1000, Level 2: 1000, Level 3: 1000, Level 4: 1000
  Other Names: 2',2'-difluorodeoxycytidine; Gem-TABS; Gemzar®

SUMMARY:
The purpose of this study is to:

Find out the largest dose of sodium bicarbonate that can be given with gemcitabine.

Determine if the combination of sodium bicarbonate and gemcitabine produces better control of pancreatic cancer than gemcitabine alone.

DETAILED DESCRIPTION:
Gemcitabine will be administered as an intravenous drip over 30 minutes at a dose of 1000 mg/m2 on days 1, 8, and 15 of each cycle followed by a 7-day treatment rest period. No treatment will be administered on the 4th week of the cycle. Each cycle is 28 days long.

Sodium bicarbonate is commercially available and supplied as tablets and water soluble powder. It is stable in solid form and does not need refrigeration. The sodium bicarbonate will be dispensed by the pharmacy in packets containing 1/3 the daily dose. The patient will be asked to dissolve the powder in water 3 times per day and consume the dose over a period of about 30 minutes.

Patients will be required to refrain from use of additional buffering agents (antacids) including sodium bicarbonate, CaCO3, and aluminum hydroxide.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed pancreatic adenocarcinoma that is metastatic or unresectable.
* Patients previously untreated with chemotherapy in the metastatic setting. Prior 5-FU or capecitabine treatment is allowed if: 1) it was given as part of a combined modality chemoradiation regimen in the adjuvant setting and; 2) no greater than 30% of bone marrow was included in the field and; 3) the treatment free interval has been ≥ 6 weeks.
* Patients must have measurable disease, defined as at least one lesion that can be measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan.
* ECOG performance status ≤2 (Karnofsky ≥60%).
* Patients must have normal organ and marrow function as defined below:

  * leukocytes ≥ 3,000/μl
  * absolute neutrophil count ≥ 1,500/μl
  * platelets ≥ 100,000/μl
  * total bilirubin ≤2.5 X institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) ≤2.5 X institutional upper limit of normal - or -
  * AST(SGOT)/ALT(SGPT) ≤5 X institutional upper limit of normal in patients with liver metastasis
  * creatinine ≤1.5 X institutional upper limit of normal and creatinine clearance > 30 ml/min (Cockcroft-Gault method)
* Has a negative serum or urine pregnancy test within 7 days prior to initiation of therapy (female patients of childbearing potential). Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential. Patients will agree to continue contraception for 30 days from the date of the last study drug administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had prior chemotherapy for pancreatic adenocarcinoma in the metastatic setting
* Patients who have received chemoradiation within the last 6 weeks prior to registration
* Patients with known allergy or severe reactions to gemcitabine
* Patients with uncontrolled hypertension and history of uncontrolled congestive heart failure
* Patients may not be receiving any other investigational agents or received investigational agents within the 28 days prior to registration.
* Patients with known brain metastases are excluded.
* Patients with active (not in remission) malignancies other than pancreatic cancer
* Pregnant women are excluded from this study because gemcitabine is a Class D agent with the potential for teratogenic or abortifacient effects.
* Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy. Therefore, HIV-positive patients receiving combination antiretroviral therapy are excluded from the study.
* Patients who require ongoing (chronic) treatment with medications, the absorption of which may be altered by NaHCO3 (benzodiazepines, flecainide, ketoconazole, lithium, iron salts, methenamine, methotrexate, quinidine, sulfa-containing antibiotics, and tetracycline), and cannot be switched to alternate medications are excluded.
* Patients who routinely use antacids including sodium bicarbonate, aluminum hydroxide, and calcium carbonate are excluded.
* Patients with a documented history of severe* COPD are excluded. *defined as GOLD stage III or greater. For patients with a documented history of COPD, pulmonary function tests to establish GOLD stage must be documented within 6 weeks prior to start of protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Establish the safety and tolerability of oral sodium bicarbonate in patients with advanced pancreatic carcinoma treated with gemcitabine | Average of 6 months

SECONDARY OUTCOMES:
Determine if oral bicarbonate improves overall survival, progression free-survival and response rate in patients with advanced pancreatic cancer | Average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Springett, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Gillies RJ, Ibrahim-Hashim A, Ordway B, Gatenby RA. Back to basic: Trials and tribulations of alkalizing agents in cancer. Front Oncol. 2022 Nov 14;12:981718. doi: 10.3389/fonc.2022.981718. eCollection 2022. PMID 36452492